CLINICAL TRIAL: NCT00461812
Title: A Single-Blind, Randomized, Positive-controlled Study to Compare Monotherapy With an Inhaled Corticosteroid (Mometasone) to Combination Therapy With an Inhaled Corticosteroid + a Long-Acting Bronchodilator (Advair) in Patients With Milder Persistent Asthma
Brief Title: A Comparison of Mometasone to Advair in Patients With Milder Persistent Asthma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: by sponsor due to failure to recruit patients who had mild persistent asthma who were not already on Advair 250/50 or 500/50.
Sponsor: Johns Hopkins University (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00001154
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mometasone (Experimental)
  Interventions: Drug: Mometasone
- Advair (Experimental)
  Interventions: Drug: Advair

INTERVENTIONS:
Drug: Mometasone
  Arms: Mometasone
Drug: Advair
  Arms: Advair

SUMMARY:
The research hypothesis for the proposed study asks the question, can Asmanex® demonstrate comparable anti-inflammatory therapeutic efficacy to the combination product, Advair® in control of mild persistent asthma?

The purpose is to demonstrate that the anti-inflammatory protection afforded by monotherapy with an inhaled steroid (Asmanex®) is comparable to combination therapy with Advair® 100/50, when measured by this standard methodology (methacholine bronchoprovocation) in subjects with mild persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* subjects 18 to 65 years of age
* a >2 year history of asthma
* FEV1 > 80% for subjects currently using Advair®.

Exclusion Criteria:

* severe asthma
* current smokers
* pregnant or breast-feeding women
* other chronic significant illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2010-01-19 (Actual); Study Completion 2010-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Creticos, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 participants were consented for this study. However, there were 23 pre-randomization screening failures. Only 10 were enrolled. The number of participants assigned/randomized to each Arm/Group is unknown.
Groups:
- All Participants: Mometasone
  or
  Advair
Period: Overall Study
Arm/Group | All Participants
Started | 10
Completed | 0
Not Completed | 10
Not completed — study terminated | 10

BASELINE CHARACTERISTICS:
Population: The number of participants assigned/randomized to each Arm/Group is unknown
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  >=18, <=16 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Assessed my Pulmonary Function Tests
Time Frame: change from baseline to study completion
Population: There is no data available for this outcome measure. The study was prematurely terminated and the PI is no longer with the institution. The information available was obtained from the IRB.
Groups:
- Mometasone: Mometasone
- Advair: Advair
Arm/Group | Mometasone | Advair
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: There is no data available for adverse events. The study was prematurely terminated and the PI is no longer with the institution. The information available was obtained from the IRB.
Groups:
- All Participants: Mometasone
  or
  Advair
  Adverse event data and the number of participants assigned to each Arm/Group is unknown because the PI left the institution and this information is unavailable
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes